CLINICAL TRIAL: NCT00172627
Title: Association and Mechanism Between Cyclooxygenase-2 and Interleukin-6 in Gastric Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Other Study IDs: 9361701204
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2005-09-15 (Estimated); Status verified 2004-12

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Time Perspective: Other

SUMMARY:
Evidence is rapidly accumulating that chronic inflammation may contribute to carcinogenesis through multiple mechanisms in a number of malignancies, including gastric carcinoma (GC). Cyclooxygenase-2 (COX-2), an inducible enzyme pivotal in the inflammatory response, converts arachidonic acid to the prostaglandins (PGs) required in initiating and maintaining reactions during the inflammatory process. Over-expression of COX-2 has been reported in a wide variety of cancers and is therefore implicated to play an important role in carcinogenesis. COX-2 can be blocked by non-steroidal anti-inflammatory drugs (NSIADs) and is currently the most studied therapeutic target of NSAIDs. Clinically, NSAIDs have long been used to treat various inflammatory or rheumatologic disorders.

Earlier clinical studies have confirmed an association between COX-2 over-expression and GC occurrence. The known mechanisms by which COX-2 promotes carcinogenesis include evasion from apoptosis, suppression of immunity, promotion of angiogenesis, and facilitation of invasiveness. However, inflammation-associated factors mediating the effects of COX-2 on carcinogenesis remain largely unknown. Interleukin-6 (IL-6) is a pro-inflammatory cytokine associated with gastritis and GC. Our earlier works has disclosed that IL-6 can promote angiogenic and anti-apoptotic ability of GC. However, the relationship between COX-2 and IL-6 in GC remains unknown.

The present study aims to investigate the clinical association between COX-2 and IL-6 in GC, to use a GC cell model for experimental study on causation and mechanism, and to verify the in vivo effect of COX-2 on IL-6 by an animal model.

We will collect 100 consecutive surgical samples of GC from the pathology archive of National Taiwan University Hospital and use immunohistochemical stain to compare protein expression in GC. The clinical study is to define certain subgroups of GC exhibiting an association between COX-2 and IL-6. In experimental study, we will clarify the causal relationship by the dose- and time-dependent experiments of COX-2 transient transfection in a GC cell line. COX-2 acts mainly via PGs, like PGE2. Therefore, we also stimulate GC cells with exogenous stimulation of PGE2 and EP receptor 1-4 agonists to determine the possible way(s) by which COX-2 induces IL-6 expression. A selective COX-2 inhibitor NS-398 and various inhibitors of PGE2 receptors are used as well to block COX-2 for determining the signaling pathway of COX-2 on IL-6. Finally, we will establish a stable COX-2 over-expressing transfectant of GC cells and its control vector transfectant for xenograft implantation study on mice. A COX-2 selective agent, celecoxib, will be administered orally to mice and tumor blocks will be harvested for determination of IL-6 expression.

The present study will provide clearer understanding of the role of COX-2 on the pro-inflammatory cytokine IL-6 in GC in both clinical and basic aspects. It might also stand for a model capable of systemically investigating the role of COX-2 on various cytokines implicated in GC.

DETAILED DESCRIPTION:
Evidence is rapidly accumulating that chronic inflammation may contribute to carcinogenesis through multiple mechanisms in a number of malignancies, including gastric carcinoma (GC). Cyclooxygenase-2 (COX-2), an inducible enzyme pivotal in the inflammatory response, converts arachidonic acid to the prostaglandins (PGs) required in initiating and maintaining reactions during the inflammatory process. Over-expression of COX-2 has been reported in a wide variety of cancers and is therefore implicated to play an important role in carcinogenesis. COX-2 can be blocked by non-steroidal anti-inflammatory drugs (NSIADs) and is currently the most studied therapeutic target of NSAIDs. Clinically, NSAIDs have long been used to treat various inflammatory or rheumatologic disorders.

Earlier clinical studies have confirmed an association between COX-2 over-expression and GC occurrence. The known mechanisms by which COX-2 promotes carcinogenesis include evasion from apoptosis, suppression of immunity, promotion of angiogenesis, and facilitation of invasiveness. However, inflammation-associated factors mediating the effects of COX-2 on carcinogenesis remain largely unknown. Interleukin-6 (IL-6) is a pro-inflammatory cytokine associated with gastritis and GC. Our earlier works has disclosed that IL-6 can promote angiogenic and anti-apoptotic ability of GC. However, the relationship between COX-2 and IL-6 in GC remains unknown.

The present study aims to investigate the clinical association between COX-2 and IL-6 in GC, to use a GC cell model for experimental study on causation and mechanism, and to verify the in vivo effect of COX-2 on IL-6 by an animal model.

We will collect 100 consecutive surgical samples of GC from the pathology archive of National Taiwan University Hospital and use immunohistochemical stain to compare protein expression in GC. The clinical study is to define certain subgroups of GC exhibiting an association between COX-2 and IL-6. In experimental study, we will clarify the causal relationship by the dose- and time-dependent experiments of COX-2 transient transfection in a GC cell line. COX-2 acts mainly via PGs, like PGE2. Therefore, we also stimulate GC cells with exogenous stimulation of PGE2 and EP receptor 1-4 agonists to determine the possible way(s) by which COX-2 induces IL-6 expression. A selective COX-2 inhibitor NS-398 and various inhibitors of PGE2 receptors are used as well to block COX-2 for determining the signaling pathway of COX-2 on IL-6. Finally, we will establish a stable COX-2 over-expressing transfectant of GC cells and its control vector transfectant for xenograft implantation study on mice. A COX-2 selective agent, celecoxib, will be administered orally to mice and tumor blocks will be harvested for determination of IL-6 expression.

The present study will provide clearer understanding of the role of COX-2 on the pro-inflammatory cytokine IL-6 in GC in both clinical and basic aspects. It might also stand for a model capable of systemically investigating the role of COX-2 on various cytokines implicated in GC.

ELIGIBILITY:
Inclusion Criteria:

* surgical samples of GC from the pathology archive of National Taiwan University Hospital

Exclusion Criteria:

* nil

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2005-01

CONTACTS AND LOCATIONS:
Overall Officials: Shih-Pei Huang, MD, Principal Investigator — Department of Internal Medicine, National Taiwan University Hospital
Locations (1):
- Shih-Pei Huang, Taipei, Taiwan